CLINICAL TRIAL: NCT04878224
Title: Junctional Zone Evaluation by 3D Ultrasound and Its Relation to Clinical Outcomes in Assisted Reproductive Technology
Brief Title: Junctional Zone and Its Relation to Outcomes in Assisted Reproductive Technology
Status: Recruiting | Type: Observational
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, Isabel Pereira, Principal investigator, Centro Hospitalar Lisboa Norte
Other Study IDs: ZJ
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Female
Keywords: infertility; ultrasound
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The junctional zone (JZ) is an internal layer of the myometrium, with unique characteristics that allow its visualization as a hypoechogenic structure in three-dimensional (3D) ultrasound.

Although traditionally evaluated by magnetic resonance imaging, 3D reconstruction offers an opportunity for reliable and easily accessible assessment. The only study that evaluated the thickness of the JZ in 3D ultrasound in the context of assisted reproductive technology (ART) found that the smaller the thickness of the JZ, the greater the rate of embryonic implantation.

This project aims to evaluate the relationship between the characteristics of the ZJ in 3D ultrasound, and the clinical outcomes of ART treatments, namely in vitro fertilization cycles, intracytoplasmic sperm injection and frozen embryo transfer (FET). Additionally, the intra and inter-observer variability of the characteristics of the JZ will be determined.

In a prospective and observational study with the inclusion of 200 cases, a 3D ultrasound will be performed on the day on which the final oocyte maturation is triggered or, on FET, on the day prior to the administration of progesterone.

The images will be evaluated independently by two observers. The principal investigator will evaluate the images in two stages.

After the quality of visualization of the JZ is classified, its thickness will be measured and described as regular, irregular or interrupted.

The volume of the ZJ will be obtained by subtracting the endometrial volume from the volume of the junctional zone and the endometrium.

These characteristics will be related to the clinical outcomes of each cycle: clinical pregnancy rate and abortion rate.

DETAILED DESCRIPTION:
After explaining the study and obtaining written consent, a 3D ultrasound will be performed for uterine evaluation, on the day of the final oocyte maturation trigger in cases of IVF / ICSI. In cases of FET, the ultrasound evaluation will be carried out on the day before the start of the luteal phase support.

All ultrasounds will be performed in a standardized manner by the same operator. With an empty bladder, in a lithotomy position, a 2D transvaginal ultrasound will be performed using a GE Voluson 730 Expert® ultrasound, with an endovaginal probe with a 4-8MHz frequency. Identification of endometriosis lesions or acquired uterine abnormalities such as leiomyomas or adenomyosis will be exclusion criteria. After evaluating the number and maximum dimension of the ovarian follicles and the endometrial thickness, the three-dimensional volume box will be placed to encompass the entire uterus in longitudinal section, with minimal inclusion of para-uterine structures. A maximum acquisition angle of 90º and maximum quality will be used. To minimize artifacts, during the acquisition both the probe and the woman must remain immobile, being asked to hold their breath. Then, a three-dimensional volume will be generated by automatic 360º rotation of the transducer. For each case, two volumes will always be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Women followed in the infertility clinic
* aged between 18 and 42 years in cycles of IVF, ICSI or endometrial preparation for frozen embryo transfer

Exclusion Criteria:

* Myomas
* adenomyosis

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women included are followed in the fertility clinic aged between 18 and 40 years in cycles of IVF, ICSI or endometrial preparation for frozen embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks
  Clinical pregnancy rate
Abortion rate | 7 weeks
  Abortion rate

SECONDARY OUTCOMES:
intra-observer variability | 2 years
  intra-observer variability
inter-observer variability | 2 years
  inter-observer variability

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Barros Pereira, M.D., Principal Investigator — Centro Hospitalar Universitário Lisboa Norte
Locations (1):
- Centro Hospitalar Universitário Lisboa Norte, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided